CLINICAL TRIAL: NCT06883734
Title: The Effect of Illness Management Skill Training Applied to Patients With Schizophrenia on Engulfment, Quality of Life and Illness Management and Recovery Levels
Brief Title: The Effect of Illness Management Skill Training Applied to Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Lok (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor-Investigator, Neslihan Lok, Prof. Dr, Study Director, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SelcukU-GUzun-002
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Schizophenia Disorder
Keywords: Schizophrenia; engulfment; quality of life; illness management; recovery; Illness Management Skills Training; psychiatric nursing
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled trial with pre-test and post-test control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group was a group of 25 people consisting of patients with schizophrenia who followed the 12-week Illness Management Skills Training.
  Interventions: Behavioral: Illness Management Skills Training
- Control (No Intervention): The control group consisted of 25 patients with schizophrenia who attended routine outpatient clinic check-ups for 12 weeks without any intervention.

INTERVENTIONS:
Behavioral: Illness Management Skills Training — In this study, in addition to routine outpatient clinic check-ups, 12 sessions of Illness Management Skills Training were applied to the intervention group of 25 patients, each in four separate groups of 6+6+6+7 patients (Group 1, Group 2, Group 3, Group 4), once a week, for 60 minutes each. The training consisted of 1) Introduction-Getting Acquainted, 2) Recovery Goals, 3) Understanding Schizophrenia-1, 4) Understanding Schizophrenia-2, 5) Stress Vulnerability Model and Coping with Stress-1, 6) Stress Vulnerability Model and Coping with Stress-2, 7) Learning About Medication, 8) Using Medication Effectively and Monitoring Treatment, 9) Coping with Persistent Symptoms, 10) Recognizing and Monitoring Warning Signs, 11) Warning Signs My Emergency Plan, and 12) Termination sessions.
  Arms: Intervention

SUMMARY:
This study was aimed to examine the effectiveness (illness management and recovery, engulfment, quality of life) of a 12-week the Illness Management Skills Training applied to patients with schizophrenia. The main questions it aims to answer are:

Hypothesis (H1-1): Illness Management Skills Training applied intervention group has lower engulfment than the control group.

Hypothesis (H1-2): Illness Management Skills Training applied intervention group has higher quality of life than the control group.

Hypothesis (H1-3): Illness Management Skills Training applied intervention group has higher illness management and recovery level than the control group.

Researchers were compared the Illness Management Skills Training to a control group (no intervention) to see if the Illness Management Skills Training works on engulfment, quality of life, illness management and recovery in patients with schizophrenia.

Participants were:

- attended the Illness Management Skills Training, one session per week for 12 weeks, 60 minutes per session, in addition to routine outpatient clinic check-ups.

DETAILED DESCRIPTION:
The study examined 110 individuals aged 18-65 who were diagnosed with schizophrenia and applied to the S.U. Faculty of Medicine Mental Health and Diseases Polyclinic in the last year, according to the inclusion-exclusion criteria. A total of 50 individuals diagnosed schizophrenia were included in the study. These individuals were randomly assigned to two groups: intervention and control. Pre-test data were collected using the "Personal Information Form", "Modified Engulfment Scale", "SF 36 Quality of Life Scale" and "Illness Management and Recovery Scale-Patient Form" from the intervention and control groups by researchers between August 2024 and February 2025 in the Group Therapy Room of the Mental Health and Diseases Polyclinic, based on self-reporting. The "Illness Management Skills Training" was applied to the intervention group in 4 groups, one session per week, for a total of 12 weeks. At the end of the Illness Management Skills Training, both the intervention and control groups were administered the "Modified Engulfment Scale", "SF 36 Quality of Life Scale" and "Illness Management and Recovery Scale-Patient Form". No intervention was applied to the control group throughout the 12-week program; the patients continued with their routine outpatient clinic check-ups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having been diagnosed with Schizophrenia for at least 6 months according to ICD-10,
* Being registered with the Selcuk University Faculty of Medical Hospital Mental Health and Diseases Polyclinic,
* Coming to the polyclinic for regular check-ups,
* Getting a mild/moderate score from the Positive and Negative Syndrome Scale (PANSS),
* Taking medication regularly,
* Being at least literate.

Exclusion Criteria:

* Having an organic mental disorder or mental retardation,
* Having a visual or hearing impairment,
* Participating in a program similar to the intervention to be implemented.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Illness management and recovery total mean score | From enrollment to the end of training at 12 weeks
  The Illness Management and Recovery Scale-Patient Form total score from the scale is 15-75. Increasing scores from the scale indicate that illness management and recovery also increase.

SECONDARY OUTCOMES:
Engulfment total mean score | From enrollment to the end of training at 12 weeks
  The score range of the Modified Engulfment Scale is 25-125. Increasing scores from the scale indicate increased engulfment .
Physical function, social function, physical role difficulty, emotional role difficulty, mental health, energy/vitality, pain and general health Physical and Mental Component Summary Scale mean scores | From enrollment to the end of training at 12 weeks
  The SF 36 Quality of Life scale evaluates quality of life through the sub-dimensions of physical function, social function, physical role difficulty, emotional role difficulty, mental health, energy/vitality, pain and general health. The scale has a physical and mental health summary scale. 0-100 points can be obtained from each sub-dimension. A score of "0" indicates poor health, while a score of 100 indicates good health, and as scores increase, the quality of life also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Lok, Prof. Dr, Study Director — Selcuk University
Locations (1):
- Selcuk University Faculty of Medical Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No